CLINICAL TRIAL: NCT03805594
Title: Immunogenic Priming With PSMA-Targeted Radioligand Therapy in Advanced Prostate Cancer: A Phase 1b Study of 177Lu-PSMA-617 in Combination With Pembrolizumab
Brief Title: 177Lu-PSMA-617 and Pembrolizumab in Treating Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Prostate Cancer Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rahul Aggarwal, Associate Clinical Professor, University of California, San Francisco
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 185511; NCI-2018-02993 (Registry Identifier: NCI Clinical Trial Reporting Program (CTRP)); R01CA229354 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Stage IV Prostate Cancer; Stage IVA Prostate Cancer; Stage IVB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A: Dosing Schedule 1 (lutetium Lu 177-PSMA-617, pembrolizumab) (Experimental): Participants receive lutetium Lu 177-PSMA-617 IV over 20-30 minutes on day 1. Beginning in cycle 2, participants receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Participants who achieve stable disease (SD) or better may receive 17 additional cycles (approximately 1 year) of pembrolizumab.
  Interventions: Drug: Lutetium Lu 177-PSMA-617; Biological: Pembrolizumab
- Part A: Dosing Schedule 2 (lutetium Lu 177-PSMA-617, pembrolizumab) (Experimental): Participants receive lutetium Lu 177-PSMA-617 IV over 20-30 minutes and pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Participants who achieve SD or better may receive 17 additional cycles (approximately 1 year) of pembrolizumab.
  Interventions: Drug: Lutetium Lu 177-PSMA-617; Biological: Pembrolizumab
- Part A: Dosing Schedule 3 (lutetium Lu 177-PSMA-617, pembrolizumab) (Experimental): Starting day -21, participants receive pembrolizumab IV over 30 minutes. Participants also receive lutetium Lu 177-PSMA-617 IV over 20-30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Participants who achieve SD or better may receive 17 additional cycles (approximately 1 year) of pembrolizumab.
  Interventions: Drug: Lutetium Lu 177-PSMA-617; Biological: Pembrolizumab
- Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (lutetium Lu 177-PSMA-617, pembrolizumab) (Experimental): Participants will receive the RP2DS determined in Part A. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Participants who achieve SD or better may receive 17 additional cycles (approximately 1 year) of pembrolizumab.
  Interventions: Drug: Lutetium Lu 177-PSMA-617; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Lutetium Lu 177-PSMA-617 — Given IV
  Other Names: 177Lu-PSMA-617; Lu177-PSMA-617
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase Ib trial studies the dose and schedule of 177Lu-PSMA-617 and pembrolizumab in treating persons with castration-resistant prostate cancer that has spread to other places in the body. 177Lu-PSMA-617 carries a radioactive component which attached to the prostate specific membrane antigen (PSMA) receptor found on tumor cells. Its radiation component destroys the tumor cell. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving 177Lu-PSMA-617 and pembrolizumab may work better at treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To determine the recommended phase 2 dose and schedule of lutetium Lu 177-PSMA-617 (177Lu-PSMA-617) in combination with pembrolizumab in participants with metastatic castration-resistant prostate carcinoma (mCRPC). (Part A)
2. To determine the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. (Part B (Dose Expansion))

SECONDARY OBJECTIVES:

1. To characterize the safety profile of the combination.
2. To determine the median duration of response by RECIST 1.1 criteria.
3. To determine the proportion of participants who experience >= 50% decline from baseline in serum prostate-specific antigen (PSA).
4. To determine the median PSA progression-free survival.
5. To determine the median time to symptomatic skeletal related event.
6. To determine the 6 month radiographic progression-free survival rate and median radiographic progression-free survival.
7. To determine the median overall survival.

CORRELATIVE OBJECTIVES:

1. To assess the lesion-specific response rate by baseline PSMA avidity on gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) positron emission tomography (PET).
2. To quantify the change from baseline in T cell repertoire, circulating T cell subsets, tumor infiltrating lymphocytes, and tumor programmed death-ligand 1 (PD-L1) expression by immunohistochemistry after one priming dose of Lu-PSMA radioligand therapy (RLT).
3. To explore the relationship between timing of the 177Lu-PSMA-617 priming dose with initiation of pembrolizumab with respect to immunologic, safety, and efficacy outcomes.
4. To descriptively characterize the patterns of uptake on 68Ga-PSMA-11 PET at the time of disease progression.
5. To explore relationship between tumor genomic profile with clinical outcomes including response rate and progression-free survival.
6. To explore the relationship between tumor dosimetry with objective response.

OUTLINE: Participants are assigned sequentially to 1 of 3 treatment schedules.

DOSING SCHEDULE 1: Participants receive lutetium Lu 177-PSMA-617 intravenously (IV) over 20-30 minutes on day 1 before beginning pembrolizumab IV over 30 minutes on day 1 in cycle 2

DOSING SCHEDULE 2: Participants receive lutetium Lu 177-PSMA-617 IV over 20-30 minutes concurrently with pembrolizumab IV over 30 minutes on day 1.

DOSING SCHEDULE 3: Starting day -21, participants receive pembrolizumab IV over 30 minutes. Participants then receive lutetium Lu 177-PSMA-617 IV over 20-30 minutes on day 1.

In all dosing schedules, treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Participants who achieve stable disease (SD) or better may receive 17 additional cycles (approximately 1 year) of pembrolizumab.

After completion of study treatment, participants are followed up at 30 days after treatment has been discontinued.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able and willing to comply with study procedures and provide signed and dated informed consent
* Histologically confirmed prostate adenocarcinoma. De novo small cell neuroendocrine prostate cancer will not be allowed due to putative lower PSMA expression in this tumor subtype. Treatment-emergent small cell neuroendocrine prostate cancer detected in metastatic tumor biopsy is not an exclusion
* A minimum of three PSMA-avid lesions on baseline 68Ga-PSMA-11 PET, with positive lesions defined as those with maximum standardized uptake value (SUVmax) values greater than liver.
* Progressive metastatic castration-resistant prostate cancer by Prostate Cancer Working Group (PCWG)3 criteria at the time of study entry
* Castrate level of serum testosterone at study entry (< 50 ng/dL). Participants without prior bilateral orchiectomy are required to remain on luteinizing hormone-releasing hormone (LHRH) analogue treatment for duration of study
* Prior progression on at least one second generation androgen signaling inhibitor including abiraterone, apalutamide, darolutamide, and/or enzalutamide
* Absolute neutrophil count > 1.5 x 10^9/L
* Hemoglobin > 9.0 g/dL
* Platelet count > 100,000/microliter
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or estimated glomerular filtration rate (GFR) > 50 ml/min by Cockcroft-Gault or 24 hour urine collection
* Total bilirubin =< 1.5 x ULN. In participants with known or suspected Gilbert's disease, direct bilirubin =< ULN
* Aspartate aminotransferase and alanine aminotransferase =< 2.5 x ULN (<= 5 x ULN in participants with liver metastases)
* No other systemic anti-cancer therapies administered other than LHRH analogue within 14 days, or 5 half-lives, whichever is shorter, prior to initiation of study treatment. Adverse events related to prior anti-cancer treatment other than LHRH analog treatment must have recovered to Grade <= 1 with the exception of any grade alopecia and grade <= 2 neuropathy.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants must use appropriate methods of contraception during study treatment and for at least 60 days after last study treatment

  * Participants who are sexually active should consider their female partner to be of childbearing potential if she has experienced menarche and is not postmenopausal (defined as amenorrhea > 24 consecutive months) or has not undergone successful surgical sterilization. Even women who use contraceptive hormones (oral, implanted, or injected), an intrauterine device, or barrier methods (diaphragms, condoms, spermicide) should be considered to be of childbearing potential
  * Participants who have undergone vasectomy themselves should also be considered to be of childbearing potential
  * Acceptable methods of contraception include continuous total abstinence, or double-barrier method of birth control (e.g. condoms used with spermicide, or condoms used with oral contraceptives). Periodic abstinence and withdrawal are not acceptable methods of contraception
* Participants must provide consent to comply to recommended radioprotection precautions during study
* Participants willing to undergo tumor biopsy and have at least one lesion safely accessible to tumor biopsy. Bone or soft tissue lesion is allowed
* Measurable disease by RECIST 1.1 criteria

Exclusion Criteria:

* Untreated brain metastases at study entry. Participants with previously treated brain metastases are eligible provided the following criteria are all met:

  * Last treatment was > 28 days prior to cycle 1 day 1 (C1D1)
  * No evidence of new/progressive brain metastases is observed on magnetic resonance imaging (MRI) obtained during screening window
  * Patient is clinically stable without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Receipt of prior PSMA-directed treatment (e.g. radiotherapy, immunotherapy, or antibody-drug conjugate)
* Prior enrollment on clinical study investigating Lu-PSMA-based radioligand therapy
* Prior treatment with radium-223 or other radioisotope for the treatment of prostate cancer
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Receipt of prior pembrolizumab or another immune checkpoint inhibitor (e.g. nivolumab, ipilimumab)
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Receipt of taxane chemotherapy applied in the castration-resistant setting. Prior receipt of taxane chemotherapy in the hormone-sensitive setting is allowed
* Grade > 2 peripheral neuropathy at the time of study entry
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) or treatment with drugs (e.g. neomercazole, carbimazole, etc.) that function to decrease the generation of thyroid hormone by a hyperfunctioning thyroid gland (e.g. in Graves? disease) is not considered a form of systemic treatment of an autoimmune disease
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a prednisone equivalent dose of > 10 mg daily or other form of immunosuppressive therapy within 7 days prior to first dose of study drug
* Has a history of (non-infectious) ≥ grade 2 pneumonitis/interstitial lung disease that required steroids within past 2 years or has current ≥ grade 1 pneumonitis/interstitial lung disease at the time of study enrollment..
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Participants who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent
* Has clinically significant cardiovascular disease including, but not limited to:

  * Uncontrolled or any New York Heart Association class 3 or 4 congestive heart failure
  * Uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months before study entry
  * Clinically significant arrhythmias not controlled by medication. Chronic rate controlled or paroxysmal atrial fibrillation/flutter is not an exclusion to study participation
* Prior external beam radiation involving >= 25% of bone marrow or within 14 days of start of protocol therapy
* Major surgery within 28 days of study treatment

  *Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) (screening not required)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection (screening not required)
* Has a known history of active Bacillus tuberculosis (TB)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Any condition that, in the opinion of the principal investigator, would impair the patient's ability to comply with study procedures
* History of bleeding diathesis and not currently on anti-coagulation therapy that cannot be safely discontinued for the tumor biopsy procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aggarwal R, Starzinski S, de Kouchkovsky I, Koshkin V, Bose R, Chou J, Desai A, Kwon D, Kaushal S, Trihy L, Rastogi M, Ippisch R, Aslam M, Friedlander T, Feng F, Oh D, Cheung A, Small E, Evans M, Fong L, Hope TA. Single-dose 177Lu-PSMA-617 followed by maintenance pembrolizumab in patients with metastatic castration-resistant prostate cancer: an open-label, dose-expansion, phase 1 trial. Lancet Oncol. 2023 Nov;24(11):1266-1276. doi: 10.1016/S1470-2045(23)00451-5. PMID 37922930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part A, three dosing schedules of priming lutetium-177 (¹⁷⁷Lu)-PSMA-617 (vipivotide tetraxetan) were assessed. Dose expansion in phase 1b (Part B) was subsequently evaluated using the recommended phase 2 dosing schedule.
Period: Overall Study
Arm/Group | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Started | 6 | 6 | 6 | 25
Completed | 6 | 6 | 6 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 25 | 43
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 1 | 1 | 1 | 2 | 5
  60-69 years old | 4 | 2 | 3 | 4 | 13
  70-79 years old | 1 | 1 | 2 | 12 | 16
  80-89 years old | 0 | 2 | 0 | 6 | 8
  90-99 years old | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 25 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 25 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 2 | 5
  White | 5 | 5 | 5 | 19 | 34
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 25 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Dose Limiting Toxicities (DLT) (Part A Only)
Description: The Recommended Phase 2 Dosing Schedule (RP2DS) (Schedule 1: a single priming dose of 177Lu-PSMA-617 (7·4 giga-becquerel (GBq) [200 millicurie (mCi)] given 28 days before pembrolizumab; Schedule 2: a single priming dose of 177Lu-PSMA-617 given concomitant with pembrolizumab; or Schedule 3: a single priming dose of 177Lu-PSMA-617 given 21 days after the start of maintenance pembrolizumab (200 mg every 3 weeks)) will be determined from the safety data as classified by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for dose-limiting toxicities, aggregate safety data and feasibility of administration. The number of dose-limiting toxicities reported by participants in Part A used to determine the RP2DS for participants enrolling under Part B will be reported by arm.
Time Frame: Up to 1 year
Population: Schedule 1, a single priming dose of 177Lu-PSMA-617 given 28 days before pembrolizumab was determined to be the RP2DS for participants enrolled under Part B
Measure: Number; unit: dose-limiting toxicities
Arm/Group | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 6 | 6 | 6
dose-limiting toxicities | 0 | 1 | 1

2. Primary Outcome: Objective Response Rate (ORR) (Part B Only)
Description: The ORR for participants in Part B is defined as the percentage of participants in Part B who obtained a confirmed diagnosis of complete response (CR) or partial response (PR), using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for the evaluation of radiographic CTs or MRIs performed during the course of the study to assess response. The ORR will be reported with a 95% confidence interval.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 25
percentage of participants | 56 [35 to 76]

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: The number of participants who reported adverse events defined by NCI CTCAE version 5.0 and attributed by the investigator to having been possibly, probably, or definitely related to study treatment will be reported.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 6 | 6 | 6 | 25
participants | 0 | 1 | 2 | 9

4. Secondary Outcome: Median Duration of Response
Description: The median duration of response in months for all participants who received at least one dose of protocol therapy (i.e., one dose of pembrolizumab or 177Lu-PSMA-617) and who also demonstrated a confirmed response of complete response (CR) or partial response (PR) per RECIST criteria from the time of first response until confirmed disease progression, death or study completion will be reported.
Time Frame: Up to 3 years
Population: Per the pre-specified statistical analysis plan outlined in the study protocol, additional efficacy endpoints other than ORR including median duration of response was planned to be analyzed in the overall study cohort (n = 43). There was no pre-specified plan to analyze efficacy outcomes by study schedule (schedule 1, 2, 3). Post-hoc determination of efficacy outcomes for schedules 1,2, 3 analyzed separately is precluded by the limited sample size on schedules 2 and 3 (n = 6 each).
Measure: Median (Full Range); unit: months
Groups:
- All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab): All participants who received any dose of lutetium Lu 177-PSMA-617 under any dosing schedule (schedule 1, 2 or 3) and given at least 1 cycle of pembrolizumab are included. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Participants who achieve stable disease (SD) or better may receive 17 additional cycles (approximately 1 year) of pembrolizumab.
Arm/Group | All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 43
months | 8.1 [6 to 10]

5. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate (PSA50)
Description: The percentage of all for all participants who received at least one dose of protocol therapy (i.e., one dose of pembrolizumab or 177Lu-PSMA-617) and who also achieved a greater than 50% decline from the time of the baseline PSA value obtained on cycle 1 day 1 (C1D1) at any point in the treatment course will be reported along with the 95% confidence interval.
Time Frame: Up to 3 years
Population: Per the pre-specified statistical analysis plan outlined in the study protocol, additional efficacy endpoints other than ORR including PSA50 was planned to be analyzed in the overall study cohort (n = 43). There was no pre-specified plan to analyze efficacy outcomes by study schedule (schedule 1, 2, 3). Post-hoc determination of efficacy outcomes for schedules 1,2, 3 analyzed separately is precluded by the limited sample size on schedules 2 and 3 (n = 6 each).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 43
percentage of participants | 44 [29 to 59]

6. Secondary Outcome: Radiographic Progression-Free Survival Rate (rPFS) at 6 Months
Description: rPFS is defined as the percentage all for all participants who received at least one dose of protocol therapy (i.e., one dose of pembrolizumab or 177Lu-PSMA-617) and who are still alive and progression-free per RECIST v1.1 and PCWG3 criteria at 6 months.
Time Frame: Up to 6 months
Population: Per the pre-specified statistical analysis plan outlined in the study protocol, additional efficacy endpoints other than ORR including rPFS at 6 months was planned to be analyzed in the overall study cohort (n = 43). There was no pre-specified plan to analyze efficacy outcomes by study schedule (schedule 1, 2, 3). Post-hoc determination of efficacy outcomes for schedules 1,2, 3 analyzed separately is precluded by the limited sample size on schedules 2 and 3 (n = 6 each).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 43
percentage of participants | 51 [35 to 67]

7. Secondary Outcome: Median PSA Progression-free Survival
Description: PSA progression-free survival for all participants who received at least one dose of protocol therapy (i.e., one dose of pembrolizumab or 177Lu-PSMA-617) will be defined using Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria as the duration in months from date of first treatment to date the participant first meets the criteria for PSA progression for clinical progression, death, or study completion, whichever occurs first. The median duration and 95% confidence interval will be reported.
Time Frame: Up to 3 years
Population: Per the pre-specified statistical analysis plan outlined in the study protocol, additional efficacy endpoints other than ORR including Median PSA progression-free survival was planned to be analyzed in overall study cohort (n = 43). There was no pre-specified plan to analyze efficacy outcomes by study schedule (schedule 1, 2, 3). Post-hoc determination of efficacy outcomes for schedules 1,2, 3 analyzed separately is precluded by the limited sample size on schedules 2 and 3 (n = 6 each).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 43
months | 6.9 [3.9 to 7.0]

8. Secondary Outcome: Median Overall Survival (OS)
Description: Median overall survival for all participants who received at least one dose of protocol therapy (i.e., one dose of pembrolizumab or 177Lu-PSMA-617) is defined as the number of months from the first date of therapy until date of death from any cause. The median number of months and 95% confidence interval will be estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Per the pre-specified statistical analysis plan outlined in the study protocol, additional efficacy endpoints other than ORR including Median Overall Survival (OS) was planned to be analyzed in overall study cohort (n = 43). There was no pre-specified plan to analyze efficacy outcomes by study schedule (schedule 1, 2, 3). Post-hoc determination of efficacy outcomes for schedules 1,2, 3 analyzed separately is precluded by the limited sample size on schedules 2 and 3 (n = 6 each).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 43
months | 28.2 [20.4 to 40.0]

9. Secondary Outcome: Median Time to Symptomatic Skeletal Related Event (SSRE)
Description: Symptomatic skeletal related event is defined as the first occurrence of one or more of the following: symptomatic fracture, surgery or radiation to bone, or spinal cord compression. The median time in months to symptomatic skeletal related event for all participants who received at least one dose of protocol therapy (i.e., one dose of pembrolizumab or 177Lu-PSMA-617) will be reported with the 95% confidence interval.
Time Frame: Up to 3 years
Population: Per the pre-specified statistical analysis plan outlined in the study protocol, additional efficacy endpoints other than ORR including median time to SSRE was planned to be analyzed in overall study cohort (n = 43). There was no pre-specified plan to analyze efficacy outcomes by study schedule (schedule 1, 2, 3). Post-hoc determination of efficacy outcomes for schedules 1, 2, 3 analyzed separately is precluded by the limited sample size on schedules 2 and 3 (n = 6 each).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants (Lutetium Lu 177-PSMA-617, Pembrolizumab)
Number analyzed (Participants) | 43
months | 24.7 [20.7 to NA] — There were insufficient number of events so the upper range of the confidence interval could not be calculated

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab) | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 4/6 | 3/6 | 4/6 | 5/25
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 1/6 | 5/25
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=6) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=6) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=6) | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=25)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Liver dysfunction
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Urosepsis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dosing Schedule 1 (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=6) | Part A: Dosing Schedule 2 (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=6) | Part A: Dosing Schedule 3 (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=6) | Part B: Recommended Phase 2 Dosing Schedule (RP2DS) (Lutetium Lu 177-PSMA-617, Pembrolizumab) (N=25)
Fatigue (General disorders) | 2 (3) | 1 (1) | 6 (10) | 20 (25)
Pain (General disorders) | 2 (2) | 1 (1) | 3 (4) | 5 (5)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localized edema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (4) | 4 (4) | 10 (11)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (4) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 6 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 3 (3) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 1 (1) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Thrombocytopenia

LIMITATIONS AND CAVEATS:
The additional efficacy endpoints including median duration of response, PSA50 response rate, rPFS rate at 6 months, median PSA progression-free survival, median OS, and median time to SSRE were planned to be analyzed in the overall study cohort (n = 43). Post-hoc determination of efficacy outcomes for schedules 1,2, 3 analyzed separately is precluded by the limited sample size of patients enrolled on schedules 2 and 3 (n = 6 each).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT03805594/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03805594/ICF_000.pdf